CLINICAL TRIAL: NCT00276198
Title: Controlled Clinical Trial to Assess the Effect of Multiple Micronutrient Supplementation (Iron, Vitamins A, C, D, Folic Acid and Zinc) on Nutritional and Health Indicators in Infants in Southern Israel.
Brief Title: Efficacy Trial to Examine Efficacy of Multimicronutrient Home Supplementation in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Naomi Amichai, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sor395705ctil
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-03

CONDITIONS: Iron Deficiency Anemia; Infectious Diseases; Undernutrition
Keywords: Clinical trial, controlled; Micronutrients; Dietary Supplementation; Infants
MeSH Terms: conditions — Anemia, Iron-Deficiency; Communicable Diseases; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Supplementation with daily sprinkle package
  Interventions: Dietary Supplement: Sprinkles
- 2 (Active Comparator): Supplementation with Iron tonic 15mg, vitamins A 300 micrograms, vitamin D 10 micrograms. According to Ministry of Health routine recommendations.
  Interventions: Dietary Supplement: Ferripel-3, Vitamins A&D drops
- 3 (No Intervention): No intervention except for checking outcomes at approprite times.

INTERVENTIONS:
Dietary Supplement: Sprinkles — Daily dosage of fat coated iron (desote fumarate) 12.5 mg, zinc 5mg, vitamin A 300 micrograms, folic acid 150 micrograms, ascorbic acid 50 mg.
  Arms: 1
Dietary Supplement: Ferripel-3, Vitamins A&D drops — Daily dosage of Iron tonic 15mg, vitamins A 300 micrograms, vitamin D 10 micrograms once a day from age 6 months up to age 12 months
  Other Names: oral drops
  Arms: 2

SUMMARY:
The objective of the program is to examine the efficacy of 6 month home micronutrient supplementation in Bedouin and Jewish children on improvements in nutritional status including measures of iron, ferritin, zinc and folic acid, and measures of growth and health parameters i.e.reported and recorded morbidity.

DETAILED DESCRIPTION:
The high level of anemia persists in Negev children despite the existence of a policy of the Ministry of Health that calls for Iron, Vitamin A and Vitamin D supplementation up to 12 months of age. In addition, other micronutrient deficiencies in this population have been described in several studies. These may be related to; low adherence with existing recommendations; need for additional micronutrients other than Iron, Vitamin A and Vitamin D; the need for a different delivery system more acceptable to mothers and infants.

We will compare in Bedouin and Jewish children separately the efficacy of daily use of Sprinkles(home Micronutrient fortification) from age 6 to 12 months in infants recruited in Maternal and Child Health clinics.

The comparison will be children recruited in clinics of comparable socioeconomic status, where current Ministry of Health recommendations (drops of iron and vitamins A plus D) are the treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 5-7 months
* Infant whose parents give their written informed consent
* Infants whose parents intend to reside within the area for at least 12 months
* Infants receiving any additional food besides breast feeding

Exclusion Criteria:

* Known or suspected haemotological disorders
* Known or suspected anemia (Hb <11 gr/dl)
* Known or suspected immunological disorders
* Known or suspected malabsorption disorders
* Enrolled or scheduled to be enrolled in another clinical trial

Ages: 5 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 771 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Haemotological parameters (haemoglobin, transferrin saturation, and ferritin) | 12, 18 and 24 months
Micronutrient status (Iron, Zinc and B12 and Folic acid level) | 12, 18 months
Incidence of infectious diseases total morbidity (IDTM) due to respiratory tract infections, diarrhea, sepsis, otitis media, cutaneous infections, fever) and all illnesses (ACTM) | 12, 18, 24 months
Health Care Services use (primary care clinics visits, emergency room visits, hospitalizations | 24 months

SECONDARY OUTCOMES:
Reported morbidity due to infectious diseases (lower respiratory tract infections, diarrhea, sepsis, otitis media, cutaneous infections, fever) | 12, 18, 24 months
Growth parameters (WAZ, HAZ, WHZ) | 12, 18, 24 months
Safety, diarrhea, constipation, color, smell and form of stool changes. Any other adverse events. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Drora Fraser, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ministry of Health, Beersheba, Israel

REFERENCES:
- [Background] Fraser D, Shahar D, Shai I, Vardi H, Bilenko N. Negev nutritional studies: nutritional deficiencies in young and elderly populations. Public Health Rev. 2000;28(1-4):31-46. PMID 11411276
- See also: The site that describes the intervention treatment — http://sghi.org/about_sprinkles/index.html